CLINICAL TRIAL: NCT05704699
Title: Effect of Early Time Restricted Eating and Brief Intense Stair Climbing on Body Composition
Brief Title: Effect of Early Eating and Stair Climbing on Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Dr. Peter Lemon, Western University, Canada
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122046
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: eTRE (Early Time Restricted Eating); eTRE With BISC (Brief Intense Stair Climbing)
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTRE (Experimental): participants allocated to this group are required to consume food during 0800h and 1600h.
  Interventions: Behavioral: eTRE
- eTRE with BISC (Active Comparator): participants allocated to this group are required to consume food during 0800h and 1600h as well as complete 3 sessions of BISC per week.
  Interventions: Behavioral: eTRE with BISC

INTERVENTIONS:
Behavioral: eTRE — eating between 0800h and 1600h daily
  Arms: eTRE
Behavioral: eTRE with BISC — eating between 0800h and 1600h daily and completing 3 sessions of BISC per week of study duration
  Arms: eTRE with BISC

SUMMARY:
To our knowledge, as of this day there are only four studies which examined the effects of eTRE with a duration of 12 weeks. There are no studies that examined this phenomenon beyond 12 weeks, one study that lasted five weeks and four studies that lasted 4 weeks or less, some even days. The four studies that lasted 12 weeks in duration all have opportunities to improve upon, which will be discussed here. The first study performed by Gabel et al., focused primarily on measuring body weight, not body composition in older adults. The eating window also began later in the morning at 1000h and finished at 1800h. There also was no restriction on participants consuming caffeine during the fasting window. The second study conducted by Gasmi et al., was focused on strictly older male participants that were active and healthy, again, without measuring body composition. The third study conducted by Wilkinson et al., did not measure body composition and the eating window lasted 10 hours instead of 8. The fourth study performed by Chow et al., examined eTRE with adults aged 45+/-12 years old and did not mention any exclusion criteria based upon physical activity levels or restrictions on caffeine/artificial sweetener intake during the fasting window. Furthermore, none of the studies mentioned above examined eTRE against eTRE with Brief Intense Stair Climbing (BISC) directly. We believe that the proposed study will address the concerns mentioned previously and further knowledge associated with eTRE.

ELIGIBILITY:
Inclusion Criteria:

* sedentary- lightly physically active (<7,500 steps daily)
* BMI > 25 • 18-39 years old

Exclusion Criteria:

* Have diabetes (self-reported)

  * Have history of smoking (self-reported)
  * Have history of cardiovascular disease (self-reported)
  * Have BMI of <24.9
* Are pregnant or become pregnant during the study (self-reported)
* Take medication for weight loss (self-reported)
* Physical activity level > 7500 steps/day
* Unstable weight for 3 months prior to commencement of study (>4kg weight loss/gain) • Employed in a shift work position

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Composition | less than 5 mins
  fat mass vs. fat-free mass via BodPod

SECONDARY OUTCOMES:
upper body strength test | < 15 mins
  3-rep max bench press
lower body strength test | < 15 mins
  3-rep max leg press
health related quality of life questionnaire | < 10 mins
  subjective feelings of well-being per participant

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Nutrition Laboratory, Western University, London, Ontario, Canada